CLINICAL TRIAL: NCT02960490
Title: A Phase 2 Study of E6011 in Subjects With Rheumatoid Arthritis Inadequately Responding to Biologics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E6011-J081-202
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis
Keywords: E6011; rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- E6011 400 mg/E6011 200 mg (Experimental): In the Treatment Phase (24 weeks), participants will receive E6011 400 milligrams (mg) at Weeks 0, 1, and 2, and then every 2 weeks subsequently until Week 10, and will then receive E6011 200 mg every 2 weeks between Weeks 12 and 22 in a double-blind manner. Participants who complete evaluations at Week 24 of the Treatment Phase will enter the Extension Phase (conducted up to Week 104 from the start of the study treatment), in which they will receive open-label E6011 200 mg every 2 weeks until Week 102.
  Interventions: Drug: E6011
- E6011 400 mg/E6011 400 mg (Experimental): In the Treatment Phase (24 weeks), participants will receive E6011 400 mg at Weeks 0, 1, and 2, and then every 2 weeks subsequently until Week 10, and will then receive E6011 400 mg every 2 weeks between Weeks 12 and 22 in a double-blind manner. Participants who complete evaluations at Week 24 of the Treatment Phase will enter the Extension Phase (conducted up to Week 104 from the start of the study treatment), in which they will receive open-label E6011 200 mg every 2 weeks until Week 102.
  Interventions: Drug: E6011
- Placebo/E6011 200 mg (Experimental): In the Treatment Phase (24 weeks), participants will receive placebo at Weeks 0, 1, and 2, and then every 2 weeks subsequently until Week 10, and will then receive E6011 200 mg every 2 weeks between Weeks 12 and 22 in a double-blind manner. Participants who complete evaluations at Week 24 of the Treatment Phase will enter the Extension Phase (conducted up to Week 104 from the start of the study treatment), in which they will receive open-label E6011 200 mg every 2 weeks until Week 102.
  Interventions: Drug: E6011; Drug: Placebo
- Placebo/E6011 400 mg (Experimental): In the Treatment Phase (24 weeks), participants will receive placebo at Weeks 0, 1, and 2, and then every 2 weeks subsequently until Week 10, and will then receive E6011 400 mg every 2 weeks between Weeks 12 and 22 in a double-blind manner. Participants who complete evaluations at Week 24 of the Treatment Phase will enter the Extension Phase (conducted up to Week 104 from the start of the study treatment), in which they will receive open-label E6011 200 mg every 2 weeks until Week 102.
  Interventions: Drug: E6011; Drug: Placebo

INTERVENTIONS:
Drug: E6011 — subcutaneous administration
Drug: Placebo — subcutaneous administration
  Arms: Placebo/E6011 200 mg; Placebo/E6011 400 mg

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled, parallel-group comparison study in rheumatoid arthritis participants inadequately responding to biologics.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and <75 years old at the time of informed consent
* Diagnosed with rheumatoid arthritis (RA) under the 1987 American College of Rheumatology (ACR) or 2010 ACR/European League Against Rheumatism (EULAR) criteria ≥12 weeks before informed consent
* Received biologics treatment under approved dosage and administration for ≥12 weeks but discontinued it before screening because of inadequate response
* History of biologics treatment should be limited to 2 agents among adalimumab, infliximab, golimumab, certolizumab pegol, etanercept, tocilizumab, and abatacept (including biosimilars)
* Presented ≥6 tender joints (out of 68 joints) and ≥6 swollen joints (out of 66 joints) in the Screening and Observation Phases
* Can continue stable dose regimen of methotrexate at 6 to 16 milligrams (mg)/week from 4 weeks before starting the study treatment until completion of the Extension Phase (or until study discontinuation)
* C-reactive protein (CRP) level ≥0.6 mg/deciliter (dL) or erythrocyte sedimentation rate (ESR) ≥28 millimeters per hour (mm/hr) in the Screening Phase
* Weighs ≥30 kilograms (kg) and ≤100 kg in the Screening Phase
* Has voluntarily consented, in writing, to participate in this study. If a participant is below the age of 20, also consented, in writing by a legally acceptable representative
* Has been thoroughly briefed on the conditions for participation in the study, is able to understand, and is willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Any history or complication of inflammatory arthritic disorder other than RA or Sjogren's syndrome
* Meets the ACR 1991 Revised Criteria for the Classification of Global Functional Status in RA Class IV in the Screening Phase
* Received immunoglobulin preparations or blood products within 24 weeks before starting the study treatment
* Received a live vaccine within 12 weeks before starting the study treatment, or is planning to receive
* Evidence of clinically significant disease (e.g., cardiac, respiratory, gastrointestinal, or renal disease) that could affect the participant's safety or interfere with the study assessments in the opinion of the investigator or subinvestigator
* Complication of uncontrolled disorders such as acute cardiac infarction, unstable angina, brain infarct, or symptomatic intracerebral hemorrhage
* History of severe allergy (shock or anaphylactoid symptoms)
* History or current clinical condition of malignant tumor, lymphoma, leukemia, or lymphoproliferative disease, except for skin carcinoma (epithelial carcinoma or basal cell carcinoma) and cervix carcinoma which has completely excised and without metastasis or recurrence for more than 5 years before informed consent
* Immunodeficiency or history of human immunodeficiency virus (HIV) infection
* Infection requiring hospitalization or intravenous administration of antibiotics or disease requiring administration of antivirus drugs (e.g., herpes zoster) within 4 weeks before starting the study treatment
* History of tuberculosis or current complication of active tuberculosis
* History of clinically important vasculitis
* Tested positive for any of the following in the Screening Phase: HIV, hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B virus core antibody (HBc antibody), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C virus antibody (HCV antibody), human T-lymphotrophic virus Type I antibody (HTLV-1 antibody), or syphilis
* Positive in tuberculosis test (QuantiFERON Tuberculosis Gold Test or T-SPOT Tuberculosis Test) in the Screening Phase
* Findings indicating a history of tuberculosis on chest x-ray in the Screening Phase
* Neurological findings such as paralysis, visual impairment, or language disorder in the Screening Phase
* Demonstrated prolonged QTcF (Fridericia's Correction Formula) interval (>450 milliseconds [ms]) in repeated electrocardiogram examinations
* Females of childbearing potential who have a positive pregnancy test in the Screening or Observation Phase or are breastfeeding
* Females of childbearing potential who:

  * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period or for 28 days after study drug discontinuation
  * Are currently abstinent, and do not agree to use a double-barrier method (as described above) or refrain from being sexually active during the study period or for 28 days after study drug discontinuation
  * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 28 days after study drug discontinuation.

(NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]).

* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period or for 28 days after study drug discontinuation). No sperm donation is allowed during the study period or for 28 days after study drug discontinuation.
* Scheduled for surgery during the study
* Currently enrolled in another clinical study or used any investigational drug or device within 28 days (or 5× the half-life, whichever is longer) before informed consent
* Has been treated with E6011 or any biologics for use in RA that has not been approved
* Use of a psychotropic agent as recreational purpose other than therapeutic purpose
* Any history of a medical condition or a concomitant medical condition that in the opinion of the investigator or subinvestigator would compromise the participant's ability to safely complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-11-26 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- Japan (45):
  - Eisai Trial Site #1, Yotsukaidō, Chiba
  - Eisai Trial Site #1, Matsuyama, Ehime
  - Eisai Trial Site #1, Kitakyushu, Fukuoka
  - Eisai Trial Site #1, Takasaki, Gunma
  - Eisai Trial Site #2, Takasaki, Gunma
  - Eisai Trial Site #1, Asahikawa, Hokkaido
  - Eisai Trial Site #1, Sapporo, Hokkaido
  - Eisai Trial Site #2, Sapporo, Hokkaido
  - Eisai Trial Site #3, Sapporo, Hokkaido
  - Eisai Trial Site #1, Katō, Hyōgo
  - Eisai Trial Site #1, Ono, Hyōgo
  - Eisai Trial Site #1, Tsukuba, Ibaraki
  - Eisai Trial Site #1, Sagamihara, Kanagawa
  - Eisai Trial Site #1, Yokohama, Kanagawa
  - Eisai Trial Site #1, Sasebo, Nagasaki
  - Eisai Trial Site #1, Tomigusuku, Okinawa
  - Eisai Trial Site #1, Kawachi-Nagano, Osaka
  - Eisai Trial Site #1, Kawagoe, Saitama
  - Eisai Trial Site #1, Kawaguchi, Saitama
  - Eisai Trial Site #1, Tokorozawa, Saitama
  - Eisai Trial Site #1, Hamamatsu, Shizuoka
  - Eisai Trial Site #1, Shimotsuke, Tochigi
  - Eisai Trial Site #1, Chūō, Tokyo
  - Eisai Trial Site #1, Fuchū, Tokyo
  - Eisai Trial Site #1, Meguro-ku, Tokyo
  - Eisai Trial Site #1, Ōta-ku, Tokyo
  - Eisai Trial Site #1, Setagaya City, Tokyo
  - Eisai Trial Site #1, Shinjuku, Tokyo
  - Eisai Trial Site #2, Shinjuku, Tokyo
  - Eisai Trial Site #1, Takaoka, Toyama
  - Eisai Trial Site #1, Chiba
  - Eisai Trial Site #1, Fukui
  - Eisai Trial Site #2, Fukuoka
  - Eisai Trial Site #3, Fukuoka
  - Eisai Trial Site #4, Fukuoka
  - Eisai Trial Site #5, Fukuoka
  - Eisai Trial Site #1, Hiroshima
  - Eisai Trial Site #1, Kagoshima
  - Eisai Trial Site #1, Kochi
  - Eisai Trial Site #1, Kyoto
  - Eisai Trial Site #1, Nagasaki
  - Eisai Trial Site #2, Nagasaki
  - Eisai Trial Site #3, Nagasaki
  - Eisai Trial Site #1, Ōita
  - Eisai Trial Site #1, Toyama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 46 investigative sites in Japan from 26 November 2016 to 25 November 2019.
Pre-assignment Details: A total of 93 participants were screened, of which 66 were randomized to receive study treatment. This study has a Core Treatment Phase (Treatment Phase: 12 Weeks; Entire Treatment Phase [Re-randomized Participants]: 12 Weeks) and an Extension Phase: 80 Weeks.
Groups:
- Core Treatment Phase: Placebo: During the Core Treatment Phase, participants received E6011-matched placebo, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 10.
- Core Treatment Phase: E6011 400 mg: During the Core Treatment Phase, participants received E6011 400 milligram (mg), infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 10.
- Core Treatment Phase: Placebo Then E6011 200 mg: Participants who received Placebo and completed Week 10 evaluations were re-randomized at Week 12 in the Core Treatment Phase to receive E6011 200 mg, infusion, subcutaneously every 2 weeks between Weeks 12 and 22. Participants who completed evaluations at Week 24 of the Core Treatment Phase entered the Extension Phase.
- Core Treatment Phase: Placebo Then E6011 400 mg: Participants who received Placebo and completed Week 10 evaluations were re-randomized at Week 12 in the Core Treatment Phase to receive E6011 400 mg, infusion, subcutaneously every 2 weeks between Weeks 12 and 22. Participants who completed evaluations at Week 24 of the Core Treatment Phase entered the Extension Phase.
- Core Treatment Phase: E6011 400 mg Then E6011 200 mg: Participants who received E6011 400 mg and completed Week 10 evaluations were re-randomized at Week 12 in the Core Treatment Phase to receive E6011 200 mg, infusion, subcutaneously every 2 weeks between Weeks 12 and 22. Participants who completed evaluations at Week 24 of the Core Treatment Phase entered the Extension Phase.
- Core Treatment Phase: E6011 400 mg Then E6011 400 mg: Participants who received E6011 400 mg and completed Week 10 evaluations were re-randomized at Week 12 in the Core Treatment Phase to receive E6011 400 mg, infusion, subcutaneously every 2 weeks between Weeks 12 and 22. Participants who completed evaluations at Week 24 of the Core Treatment Phase entered the Extension Phase.
- Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg: Participants who received Placebo up to Week 10 followed by E6011 200 mg from Weeks 12 to 22 during the Core Treatment Phase continued receiving E6011 200 mg, infusion, subcutaneously every 2 weeks up to Week 102 in the Extension Phase.
- Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg: Participants who received Placebo up to Week 10 followed by E6011 400 mg from Weeks 12 to 22 during the Core Treatment Phase continued receiving E6011 200 mg, infusion, subcutaneously every 2 weeks up to Week 102 in the Extension Phase.
- Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg: Participants who received E6011 400 mg up to Week 10 followed by E6011 200 mg from Weeks 12 to 22 during the Core Treatment Phase continued receiving E6011 200 mg, infusion, subcutaneously every 2 weeks up to Week 102 in the Extension Phase.
- Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg: Participants who received E6011 400 mg up to Week 10 followed by E6011 400 mg from Weeks 12 to 22 during the Core Treatment Phase continued receiving E6011 200 mg, infusion, subcutaneously every 2 weeks up to Week 102 in the Extension Phase.
Period: Treatment Phase(Double-blind): 12 Weeks
Arm/Group | Core Treatment Phase: Placebo | Core Treatment Phase: E6011 400 mg | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Started | 34 | 32 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 33 | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Full Analysis Set (FAS) | 33 | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Safety Analysis Set (SAS) | 33 | 31 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 29 | 26 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not treated | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Re-randomized Participants: 12 Weeks
Arm/Group | Core Treatment Phase: Placebo | Core Treatment Phase: E6011 400 mg | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Started | 0 | 0 | 15 | 14 | 14 | 12 | 0 | 0 | 0 | 0
Treated | 0 | 0 | 15 | 14 | 14 | 12 | 0 | 0 | 0 | 0
FAS | 0 | 0 | 15 | 14 | 14 | 12 | 0 | 0 | 0 | 0
SAS | 0 | 0 | 15 | 14 | 14 | 12 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 13 | 12 | 13 | 10 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Phase(Open-label): 80 Weeks
Arm/Group | Core Treatment Phase: Placebo | Core Treatment Phase: E6011 400 mg | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 11 (One Participant who completed Core Treatment Phase (Placebo Then E6011 400 mg arm) had inadequate therapeutic effect at Week 24, hence did not started Extension phase.) | 13 | 10
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
FAS | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
SAS | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 5 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 4 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 7
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The FAS was the group of randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement.
Groups:
- Core Treatment Phase: Placebo: During the Core Treatment Phase, participants received E6011-matched placebo, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 10. Participants who continued the study beyond Week 12 in the Core Treatment Phase (Placebo) received E6011 200 mg or 400 mg, infusion, subcutaneously every 2 weeks between weeks 12 and 22. Participants who completed evaluations at Week 24 of the Core Treatment Phase entered the Extension Phase.
- Core Treatment Phase: E6011 400 mg: During the Core Treatment Phase, participants received E6011 400 mg, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 10. Participants who continued the study beyond Week 12 in the Core Treatment Phase (E6011 400 mg) received E6011 200 mg or 400 mg, infusion, subcutaneously every 2 weeks between weeks 12 and 22. Participants who completed evaluations at Week 24 of the Core Treatment Phase entered the Extension Phase.
- Total: Total of all reporting groups
Arm/Group | Core Treatment Phase: Placebo | Core Treatment Phase: E6011 400 mg | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (10.64) | 53.5 (11.30) | 51.5 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 5 | 9 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 33 | 31 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 33 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Core Treatment Phase: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 12 Based on Non-responder Imputation (NRI)
Description: The ACR20 response was defined as if the following 3 criteria (ACR components) were met: Greater than or equal to (>=) 20 percent (%) reduction from baseline in the tender joint count (TJC) in 68 joints (TJC68); >=20% reduction from baseline in the swollen joint count (SJC) in 66 joints (SJC66); >=20% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (visual analog scale [VAS]), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), Health Assessment Questionnaire disability index (HAQ-DI), and C-reactive protein (CRP).
Time Frame: Week 12
Population: FAS included all randomized participants who received at least 1 dose of study drug and had at least 1 postdose primary efficacy measurement. Non-responders (due to early discontinuation or other reasons were considered non-responders) imputation was applied for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Core Treatment Phase: E6011 400 mg: During the Core Treatment Phase, participants received E6011 400 mg, infusion, subcutaneously, at Weeks 0, 1, and 2 and then every 2 weeks up to Week 10.
Arm/Group | Core Treatment Phase: Placebo | Core Treatment Phase: E6011 400 mg
Number analyzed (Participants) | 33 | 31
percentage of participants | 27.3 [12.08 to 42.47] | 22.6 [7.86 to 37.30]
Statistical Analysis 1: Comparison: Core Treatment Phase: Placebo vs Core Treatment Phase: E6011 400 mg; Test type: Superiority; p = 0.621, Regression, Logistic; Difference from Placebo = -4.7, 95% CI 2-sided [-25.85 to 16.46]

2. Secondary Outcome: Percentage of Participants Who Achieved an ACR20 Response at Weeks 2, 4, 8, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72 Based on NRI
Description: The ACR20 response was defined as if the following 3 criteria (ACR components) were met: >=20% reduction from baseline in the TJC in 68 joints (TJC68); >=20% reduction from baseline in the SJC in 66 joints (SJC66); >=20% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (VAS), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), HAQ-DI, and CRP. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: Core Treatment Phase: Weeks 2, 4, 8, 16, 20, 24; Extension Phase: Weeks 2, 4, 8, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72
Population: FAS included all re-randomized participants who received at least 1 dose of study drug, and had at least 1 primary efficacy measurement. Here number analyzed "n" were the participants who were evaluable for the outcome measure for given time points. Non-responders (due to early discontinuation or other reasons were considered non-responders) imputation was applied for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
percentage of participants
  Response at Week 2 | 13.3 [0.00 to 30.54] | 7.1 [0.00 to 20.63] | 7.1 [0.00 to 20.63] | 25.0 [0.50 to 49.50] | 15.4 [0.00 to 35.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Response at Week 4 | 13.3 [0.00 to 30.54] | 28.6 [4.91 to 52.24] | 28.6 [4.91 to 52.24] | 8.3 [0.00 to 23.97] | 15.4 [0.00 to 35.00] | 27.3 [0.95 to 53.59] | 30.8 [5.68 to 55.86] | 10.0 [0.00 to 28.59]
  Response at Week 8 | 20.0 [0.00 to 40.24] | 28.6 [4.91 to 52.24] | 35.7 [10.61 to 60.81] | 25.0 [0.50 to 49.50] | 23.1 [0.17 to 45.98] | 27.3 [0.95 to 53.59] | 38.5 [12.02 to 64.91] | 30.0 [1.60 to 58.40]
  Response at Week 16 | 26.7 [4.29 to 49.05] | 28.6 [4.91 to 52.24] | 42.9 [16.93 to 68.78] | 50.0 [21.71 to 78.29] | 30.8 [5.68 to 55.86] | 36.4 [7.94 to 64.79] | 46.2 [19.05 to 73.25] | 60.0 [29.64 to 90.36]
  Response at Week 20 | 46.7 [21.42 to 71.91] | 35.7 [10.61 to 60.81] | 28.6 [4.91 to 52.24] | 50.0 [21.71 to 78.29] | 53.8 [26.75 to 80.95] | 45.5 [16.03 to 74.88] | 30.8 [5.68 to 55.86] | 50.0 [19.01 to 80.99]
  Response at Week 24 | 46.7 [21.42 to 71.91] | 28.6 [4.91 to 52.24] | 21.4 [0.00 to 42.92] | 33.3 [6.66 to 60.01] | 53.8 [26.75 to 80.95] | 36.4 [7.94 to 64.79] | 23.1 [0.17 to 45.98] | 30.0 [1.60 to 58.40]
  Response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 28 |  |  |  |  | 53.8 [26.75 to 80.95] | 54.5 [25.12 to 83.97] | 38.5 [12.02 to 64.91] | 50.0 [19.01 to 80.99]
  Response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 32 |  |  |  |  | 61.5 [35.09 to 87.98] | 36.4 [7.94 to 64.79] | 38.5 [12.02 to 64.91] | 50.0 [19.01 to 80.99]
  Response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 36 |  |  |  |  | 46.2 [19.05 to 73.25] | 36.4 [7.94 to 64.79] | 38.5 [12.02 to 64.91] | 50.0 [19.01 to 80.99]
  Response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 40 |  |  |  |  | 61.5 [35.09 to 87.98] | 36.4 [7.94 to 64.79] | 30.8 [5.68 to 55.86] | 40.0 [9.64 to 70.36]
  Response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 44 |  |  |  |  | 61.5 [35.09 to 87.98] | 45.5 [16.03 to 74.88] | 38.5 [12.02 to 64.91] | 40.0 [9.64 to 70.36]
  Response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 48 |  |  |  |  | 53.8 [26.75 to 80.95] | 54.5 [25.12 to 83.97] | 53.8 [26.75 to 80.95] | 40.0 [9.64 to 70.36]
  Response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 52 |  |  |  |  | 38.5 [12.02 to 64.91] | 45.5 [16.03 to 74.88] | 53.8 [26.75 to 80.95] | 50.0 [19.01 to 80.99]
  Response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 56 |  |  |  |  | 53.8 [26.75 to 80.95] | 27.3 [0.95 to 53.59] | 38.5 [12.02 to 64.91] | 20.0 [0.00 to 44.79]
  Response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 60 |  |  |  |  | 46.2 [19.05 to 73.25] | 18.2 [0.00 to 40.97] | 38.5 [12.02 to 64.91] | 30.0 [1.60 to 58.40]
  Response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 64 |  |  |  |  | 46.2 [19.05 to 73.25] | 27.3 [0.95 to 53.59] | 46.2 [19.05 to 73.25] | 20.0 [0.00 to 44.79]
  Response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 68 |  |  |  |  | 38.5 [12.02 to 64.91] | 27.3 [0.95 to 53.59] | 38.5 [12.02 to 64.91] | 20.0 [0.00 to 44.79]
  Response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 72 |  |  |  |  | 38.5 [12.02 to 64.91] | 45.5 [16.03 to 74.88] | 53.8 [26.75 to 80.95] | 20.0 [0.00 to 44.79]

3. Secondary Outcome: Percentage of Participants Who Achieved an ACR50 Response at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72 Based on NRI
Description: The ACR50 response was defined as if the following 3 criteria (ACR components) were met: >=50% reduction from baseline in the TJC in 68 joints (TJC68); >=50% reduction from baseline in the SJC in 66 joints (SJC66); >=50% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (VAS), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), HAQ-DI, and CRP. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: Core Treatment Phase: Weeks 2, 4, 8, 12, 16, 20 and 24; Extension Phase: Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
percentage of participants
  Response at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Response at Week 4 | 0.0 [0.00 to 0.00] | 14.3 [0.00 to 32.62] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Response at Week 8 | 0.0 [0.00 to 0.00] | 14.3 [0.00 to 32.62] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Response at Week 12 | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 7.1 [0.00 to 20.63] | 16.7 [0.00 to 37.75] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Response at Week 16 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 16.7 [0.00 to 37.75] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Response at Week 20 | 20.0 [0.00 to 40.24] | 7.1 [0.00 to 20.63] | 7.1 [0.00 to 20.63] | 16.7 [0.00 to 37.75] | 23.1 [0.17 to 45.98] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Response at Week 24 | 20.0 [0.00 to 40.24] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 16.7 [0.00 to 37.75] | 23.1 [0.17 to 45.98] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 28 |  |  |  |  | 30.8 [5.68 to 55.86] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 30.0 [1.60 to 58.40]
  Response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 32 |  |  |  |  | 15.4 [0.00 to 35.00] | 9.1 [0.00 to 26.08] | 30.8 [5.68 to 55.86] | 20.0 [0.00 to 44.79]
  Response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 36 |  |  |  |  | 23.1 [0.17 to 45.98] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 40 |  |  |  |  | 15.4 [0.00 to 35.00] | 9.1 [0.00 to 26.08] | 23.1 [0.17 to 45.98] | 20.0 [0.00 to 44.79]
  Response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 44 |  |  |  |  | 30.8 [5.68 to 55.86] | 27.3 [0.95 to 53.59] | 23.1 [0.17 to 45.98] | 10.0 [0.00 to 28.59]
  Response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 48 |  |  |  |  | 23.1 [0.17 to 45.98] | 27.3 [0.95 to 53.59] | 30.8 [5.68 to 55.86] | 20.0 [0.00 to 44.79]
  Response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 52 |  |  |  |  | 15.4 [0.00 to 35.00] | 27.3 [0.95 to 53.59] | 30.8 [5.68 to 55.86] | 10.0 [0.00 to 28.59]
  Response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 56 |  |  |  |  | 23.1 [0.17 to 45.98] | 18.2 [0.00 to 40.97] | 23.1 [0.17 to 45.98] | 10.0 [0.00 to 28.59]
  Response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 60 |  |  |  |  | 30.8 [5.68 to 55.86] | 18.2 [0.00 to 40.97] | 30.8 [5.68 to 55.86] | 20.0 [0.00 to 44.79]
  Response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 64 |  |  |  |  | 23.1 [0.17 to 45.98] | 18.2 [0.00 to 40.97] | 23.1 [0.17 to 45.98] | 10.0 [0.00 to 28.59]
  Response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 68 |  |  |  |  | 23.1 [0.17 to 45.98] | 9.1 [0.00 to 26.08] | 23.1 [0.17 to 45.98] | 10.0 [0.00 to 28.59]
  Response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 72 |  |  |  |  | 15.4 [0.00 to 35.00] | 27.3 [0.95 to 53.59] | 30.8 [5.68 to 55.86] | 10.0 [0.00 to 28.59]

4. Secondary Outcome: Percentage of Participants Who Achieved an ACR70 Response at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72 Based on NRI
Description: The ACR70 response was defined as if the following 3 criteria (ACR components) were met: >=70% reduction from baseline in the TJC in 68 joints (TJC68); >=70% reduction from baseline in the SJC in 66 joints (SJC66); >=70% reduction from baseline in at least 3 of the following 5 assessments: Physician's Global Assessment of Disease Activity (VAS), Participant's Global Assessment of Disease Activity (VAS), Participant's Assessment of Pain (VAS), HAQ-DI, and CRP. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
percentage of participants
  Response at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Response at Week 4 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Response at Week 8 | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Response at Week 12 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Response at Week 16 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Response at Week 20 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 8.3 [0.00 to 23.97] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Response at Week 24 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 28 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 32 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 0.0 [0.00 to 0.00]
  Response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 36 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 40 |  |  |  |  | 7.7 [0.00 to 22.18] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 44 |  |  |  |  | 7.7 [0.00 to 22.18] | 18.2 [0.00 to 40.97] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 48 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 52 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 56 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 60 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 64 |  |  |  |  | 7.7 [0.00 to 22.18] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 68 |  |  |  |  | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Response at Week 72 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]

5. Secondary Outcome: Change From Baseline in Tender Joint Counts (TJC) at Each Visit Based on Last Observation Carried Forward (LOCF)
Description: A total of 28 joints were examined for tenderness by applying pressure to the joint line or by moving joints through their respective ranges of motion. Joints were examined for tenderness by applying pressure to the joint line or by moving joints through their respective ranges of motion. Tender joints were marked with tick or cross in corresponding frames of the Assessment Sheet for Tender Joint Counts. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: Core Treatment Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20 and 24; Extension Phase: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68 and 72
Population: FAS included all re-randomized participants who received at least 1 dose of study drug, and had at least 1 primary efficacy measurement. Here number analyzed "n" were the participants who were evaluable for the outcome measure for given time points. LOCF imputation was applied for missing data.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
tender joints
  Baseline | 9.7 (6.88) | 11.7 (7.74) | 9.9 (4.80) | 12.8 (7.58) | 8.7 (4.85) | 11.6 (8.67) | 9.5 (4.75) | 10.3 (5.10)
  Change at Week 2 | -1.6 (3.92) | -1.3 (3.41) | -1.9 (4.48) | -4.4 (5.52) | -2.0 (4.06) | -1.3 (3.77) | -2.0 (4.65) | -3.0 (4.83)
  Change at Week 4 | -2.8 (6.07) | -2.9 (5.11) | -2.3 (5.81) | -5.1 (6.16) | -3.2 (6.48) | -3.1 (5.74) | -1.8 (5.80) | -3.9 (5.92)
  Change at Week 8 | -3.3 (5.51) | -2.9 (8.89) | -1.9 (6.18) | -5.8 (3.05) | -3.5 (5.91) | -3.8 (9.72) | -1.3 (6.06) | -5.2 (2.97)
  Change at Week 12 | -2.7 (5.59) | -2.1 (8.75) | -2.0 (6.11) | -6.2 (3.86) | -3.1 (5.92) | -3.5 (9.05) | -1.8 (6.30) | -6.1 (4.20)
  Change at Week 16 | -4.3 (6.65) | -4.1 (5.17) | -2.9 (5.73) | -7.5 (6.97) | -4.5 (7.15) | -4.8 (5.38) | -2.6 (5.84) | -6.5 (5.72)
  Change at Week 20 | -4.9 (6.06) | -4.1 (7.19) | -2.9 (6.46) | -8.2 (7.30) | -5.2 (6.48) | -4.9 (7.82) | -2.8 (6.72) | -6.3 (4.16)
  Change at Week 24 | -5.1 (5.63) | -3.7 (8.30) | -2.6 (6.06) | -7.8 (8.07) | -5.5 (5.99) | -3.9 (9.81) | -2.5 (6.29) | -6.2 (6.89)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -4.6 (6.64) | -4.5 (10.32) | -2.4 (7.54) | -4.7 (4.69)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -3.7 (7.16) | -3.9 (9.08) | -3.5 (8.42) | -5.3 (6.52)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -4.7 (7.04) | -5.0 (8.93) | -3.5 (7.61) | -4.5 (8.10)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -3.8 (7.16) | -5.1 (8.56) | -3.2 (7.72) | -4.1 (6.72)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -4.5 (7.17) | -5.5 (8.99) | -3.6 (7.89) | -4.4 (8.29)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -4.2 (7.32) | -5.5 (9.37) | -2.9 (7.71) | -2.9 (6.72)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -2.5 (6.83) | -5.8 (9.90) | -3.8 (7.93) | -4.9 (6.94)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -2.8 (6.88) | -6.3 (10.25) | -2.8 (8.00) | -4.5 (7.59)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -2.8 (6.80) | -4.5 (7.33) | -3.5 (8.12) | -4.5 (7.74)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -2.6 (6.79) | -2.6 (6.41) | -4.1 (8.27) | -4.4 (7.52)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -2.8 (6.72) | -4.6 (8.03) | -2.9 (8.20) | -4.1 (7.05)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -2.8 (6.65) | -5.5 (9.03) | -3.5 (8.33) | -4.1 (7.46)

6. Secondary Outcome: Change From Baseline in Swollen Joint Counts (SJC) at Each Visit Based on LOCF
Description: A total of 28 joints were examined for swollen joints. Swollen joints were marked with open circles in corresponding frames of the Assessment Sheet for Swollen Joint Counts. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
swollen joints
  Baseline | 7.1 (2.91) | 9.5 (6.14) | 8.9 (3.47) | 8.8 (4.39) | 7.0 (2.97) | 9.5 (6.98) | 9.2 (3.51) | 7.6 (3.37)
  Change at Week 2 | -2.7 (2.99) | -2.6 (2.31) | -2.0 (2.86) | -3.3 (4.69) | -2.7 (3.17) | -2.7 (2.57) | -2.2 (2.91) | -2.6 (4.77)
  Change at Week 4 | -2.3 (3.73) | -3.7 (3.95) | -1.8 (3.60) | -3.9 (4.14) | -2.4 (3.75) | -3.5 (4.44) | -1.9 (3.71) | -3.9 (4.48)
  Change at Week 8 | -3.3 (3.33) | -4.8 (6.38) | -0.8 (4.54) | -4.8 (4.15) | -3.5 (3.33) | -5.1 (7.20) | -0.8 (4.72) | -5.0 (4.57)
  Change at Week 12 | -2.9 (3.95) | -4.2 (6.40) | -2.5 (4.01) | -4.3 (4.61) | -3.5 (3.95) | -4.5 (7.22) | -2.8 (4.04) | -4.2 (4.83)
  Change at Week 16 | -3.2 (4.06) | -5.4 (5.45) | -1.9 (4.57) | -5.3 (4.63) | -3.5 (3.95) | -5.6 (6.17) | -1.9 (4.75) | -5.1 (4.75)
  Change at Week 20 | -3.3 (4.60) | -5.8 (6.10) | -1.4 (4.82) | -5.8 (4.34) | -3.2 (4.76) | -6.0 (6.65) | -1.4 (4.82) | -5.5 (4.22)
  Change at Week 24 | -3.9 (4.45) | -5.4 (7.26) | -0.6 (5.65) | -4.0 (3.79) | -4.4 (4.33) | -4.9 (8.97) | -0.8 (5.83) | -4.1 (4.18)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -4.1 (3.95) | -5.6 (7.85) | -1.1 (5.63) | -4.6 (2.84)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -3.7 (3.43) | -5.3 (7.99) | -1.1 (6.50) | -4.5 (5.28)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -3.7 (3.75) | -5.7 (7.67) | -1.2 (6.95) | -3.7 (6.67)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -3.5 (3.64) | -5.5 (7.94) | -2.8 (7.01) | -3.8 (6.58)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -2.5 (6.65) | -5.6 (7.84) | -1.8 (7.00) | -2.8 (6.55)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -3.5 (3.41) | -5.5 (8.18) | -2.0 (6.43) | -3.1 (5.84)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -2.4 (4.03) | -4.9 (8.58) | -1.5 (6.57) | -4.3 (6.52)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -2.8 (4.12) | -5.1 (8.70) | -2.1 (6.51) | -3.7 (6.68)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -2.8 (4.16) | -4.3 (7.93) | -2.7 (7.25) | -4.1 (6.49)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -2.5 (3.93) | -4.0 (7.89) | -1.8 (7.56) | -3.6 (6.77)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -2.8 (4.13) | -4.0 (8.31) | -1.6 (6.95) | -3.4 (6.57)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -2.7 (4.03) | -4.5 (9.11) | -2.6 (7.31) | -3.1 (6.56)

7. Secondary Outcome: Change From Baseline in Participant's Assessment of Pain Based on VAS Score at Each Visit Based on LOCF
Description: Intensity and severity of pain associated with rheumatoid arthritis (RA) were indicated by the participant on a score sheet, Pain/disease activity assessments reported by the participant, by placing a mark on a 100 millimeter (mm) horizontal VAS. Pain assessments reported by the participant, by placing a mark on a 100 mm horizontal VAS. The scale ranged from 0-100 mm, where 0 indicated no disease activity (symptom free and no arthritis symptoms) and 100 represented maximum disease activity (maximum arthritis disease activity). Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
millimeter
  Baseline | 56.7 (32.02) | 55.9 (30.33) | 56.9 (33.07) | 60.3 (20.78) | 57.5 (28.43) | 52.5 (29.96) | 54.2 (32.67) | 56.4 (18.78)
  Change at Week 2 | -5.7 (15.50) | -3.3 (15.47) | -3.3 (22.53) | -4.8 (19.07) | -7.4 (15.71) | -3.4 (17.57) | -3.0 (23.42) | -1.9 (19.67)
  Change at Week 4 | -9.8 (16.50) | -13.4 (26.58) | -8.4 (21.23) | -6.3 (17.61) | -11.2 (17.32) | -12.0 (27.40) | -7.5 (21.82) | -8.8 (18.18)
  Change at Week 8 | -13.9 (18.95) | -14.2 (30.92) | -9.6 (21.94) | -12.6 (14.88) | -14.7 (19.04) | -12.8 (34.33) | -7.5 (21.19) | -14.1 (15.81)
  Change at Week 12 | -8.5 (25.01) | -8.0 (24.10) | -15.1 (18.89) | -16.8 (20.23) | -9.5 (23.09) | -7.6 (26.27) | -14.2 (19.33) | -16.4 (18.84)
  Change at Week 16 | -15.7 (23.03) | -9.8 (18.35) | -18.5 (22.70) | -15.9 (14.77) | -16.4 (24.02) | -11.4 (20.57) | -17.8 (23.49) | -14.7 (12.96)
  Change at Week 20 | -18.4 (28.02) | -9.2 (15.57) | -14.7 (23.67) | -17.7 (16.88) | -22.8 (23.35) | -9.5 (16.32) | -15.0 (24.61) | -14.2 (13.38)
  Change at Week 24 | -17.4 (27.91) | -8.4 (18.57) | -20.0 (28.15) | -14.9 (14.69) | -21.6 (23.42) | -9.9 (20.54) | -20.7 (29.18) | -12.9 (14.65)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -21.0 (31.09) | -11.4 (21.87) | -21.8 (22.14) | -13.3 (21.07)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -18.5 (28.19) | -10.2 (22.65) | -18.9 (31.30) | -13.9 (18.53)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -19.4 (30.09) | -14.1 (29.22) | -16.0 (31.43) | -14.1 (17.95)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -19.5 (25.19) | -10.5 (28.04) | -16.6 (27.97) | -10.3 (17.97)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -22.6 (28.54) | -15.1 (35.60) | -18.2 (29.42) | -8.3 (16.59)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -20.3 (29.20) | -13.9 (34.19) | -20.8 (30.17) | -10.1 (20.25)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -21.5 (26.83) | -13.8 (36.26) | -20.8 (30.07) | -8.8 (17.57)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -23.5 (26.93) | -14.2 (33.99) | -17.3 (28.80) | -8.3 (17.86)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -21.3 (31.66) | -8.2 (27.93) | -16.6 (27.52) | -7.3 (17.09)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -19.9 (27.82) | -7.1 (24.97) | -19.1 (31.38) | -5.6 (17.02)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -21.3 (29.91) | -6.5 (21.29) | -17.7 (31.37) | -5.5 (15.59)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -22.5 (26.09) | -10.5 (26.79) | -18.9 (33.97) | -4.0 (14.57)

8. Secondary Outcome: Change From Baseline in Participant's Global Assessment of Disease Activity Based on VAS Score at Each Visit Based on LOCF
Description: Participants were evaluated on their disease activity of RA, and entered the result on the score sheet, disease activity assessments reported by the participant, by placing a mark on a 100 mm horizontal VAS. The scale ranged from 0-100 mm, where 0 indicated no disease activity (symptom free and no arthritis symptoms) and 100 represented maximum disease activity (maximum arthritis disease activity). Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
millimeter
  Baseline | 56.2 (31.20) | 54.9 (32.83) | 55.6 (34.74) | 57.7 (20.12) | 57.2 (27.56) | 51.0 (32.93) | 52.3 (33.74) | 53.9 (18.43)
  Change at Week 2 | -1.4 (10.52) | -4.1 (13.20) | -4.6 (20.66) | -4.7 (14.21) | -2.6 (10.59) | -4.2 (14.70) | -3.6 (21.18) | -2.7 (14.71)
  Change at Week 4 | -8.1 (16.76) | -12.7 (25.46) | -7.4 (24.36) | -3.9 (14.72) | -9.3 (17.76) | -11.5 (25.73) | -5.5 (24.34) | -7.0 (13.75)
  Change at Week 8 | -11.5 (19.27) | -13.4 (29.22) | -8.9 (24.79) | -14.8 (16.50) | -12.3 (19.83) | -11.6 (32.31) | -6.0 (23.28) | -13.4 (15.37)
  Change at Week 12 | -7.2 (25.53) | -6.9 (23.69) | -13.1 (22.86) | -13.1 (20.03) | -8.5 (24.24) | -5.8 (24.73) | -12.2 (23.48) | -13.9 (18.33)
  Change at Week 16 | -15.0 (25.59) | -7.4 (18.94) | -14.1 (24.07) | -13.5 (17.73) | -16.2 (27.05) | -9.5 (20.91) | -13.6 (24.99) | -13.0 (18.05)
  Change at Week 20 | -16.7 (27.33) | -8.4 (14.28) | -12.7 (26.93) | -16.8 (20.74) | -20.9 (24.16) | -9.4 (15.21) | -12.4 (28.00) | -13.6 (19.38)
  Change at Week 24 | -15.9 (27.17) | -8.8 (16.43) | -16.3 (27.10) | -12.3 (13.50) | -20.0 (24.13) | -10.8 (17.92) | -16.2 (28.20) | -11.3 (14.59)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -19.2 (27.12) | -13.7 (22.84) | -17.7 (21.66) | -11.2 (25.45)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -17.4 (23.95) | -10.5 (24.46) | -14.2 (24.86) | -10.3 (21.95)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -18.7 (27.02) | -17.4 (31.23) | -9.5 (25.94) | -10.9 (21.74)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -17.7 (22.48) | -13.3 (26.52) | -14.5 (24.66) | -7.7 (18.61)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -22.9 (27.86) | -16.5 (32.23) | -14.5 (25.67) | -5.2 (17.14)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -22.9 (27.38) | -17.2 (35.22) | -16.5 (26.51) | -5.3 (21.65)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -20.9 (24.80) | -18.3 (35.75) | -16.6 (25.83) | -4.0 (19.56)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -23.5 (25.13) | -16.6 (34.47) | -13.2 (23.44) | -3.5 (19.43)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -21.4 (29.91) | -11.2 (27.25) | -12.8 (23.57) | -4.7 (20.23)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -20.5 (26.49) | -9.2 (27.18) | -14.1 (25.89) | -2.3 (19.11)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -20.7 (28.39) | -8.2 (22.01) | -13.5 (24.90) | -0.9 (17.86)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -21.9 (24.06) | -13.5 (27.56) | -14.2 (27.03) | 0.2 (16.61)

9. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity Scale Based on VAS Score at Each Visit Based on LOCF
Description: The Physician's Global Assessment of Disease Activity was recorded using the 100 mm horizontal VAS. Physician rated participant's RA disease activity on a scale ranged from 0-100 mm, where 0 indicated no disease activity (no arthritis) and 100 represented maximum disease activity (maximum arthritis). Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
millimeter
  Baseline | 63.3 (29.63) | 57.9 (22.02) | 62.4 (19.41) | 54.0 (27.28) | 60.8 (30.56) | 56.4 (22.41) | 60.5 (18.80) | 49.6 (27.15)
  Change at Week 2 | -16.8 (16.83) | -13.6 (17.95) | -13.3 (23.08) | -8.1 (18.53) | -15.6 (17.52) | -16.8 (17.66) | -13.9 (23.89) | -6.6 (20.13)
  Change at Week 4 | -20.7 (13.62) | -16.8 (19.68) | -17.8 (27.46) | -10.1 (16.68) | -18.2 (12.60) | -16.7 (16.88) | -17.7 (28.58) | -12.7 (17.13)
  Change at Week 8 | -23.8 (26.32) | -17.6 (21.57) | -19.6 (27.81) | -13.8 (18.01) | -17.7 (22.40) | -17.7 (20.60) | -20.3 (28.83) | -14.6 (19.79)
  Change at Week 12 | -23.3 (26.50) | -9.4 (21.99) | -19.0 (30.18) | -14.7 (21.15) | -20.5 (24.71) | -11.5 (20.62) | -20.8 (30.65) | -17.2 (22.32)
  Change at Week 16 | -28.4 (30.15) | -19.7 (20.22) | -23.4 (29.34) | -14.5 (23.89) | -23.6 (29.57) | -23.1 (20.53) | -24.5 (30.19) | -16.7 (25.66)
  Change at Week 20 | -28.9 (25.67) | -24.3 (22.97) | -20.6 (27.81) | -19.1 (20.38) | -25.9 (25.94) | -30.2 (20.74) | -21.7 (28.61) | -19.7 (19.93)
  Change at Week 24 | -36.7 (30.38) | -18.3 (21.35) | -17.6 (26.03) | -10.0 (23.18) | -34.8 (32.06) | -22.6 (20.34) | -18.5 (26.87) | -8.9 (23.36)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -35.1 (36.51) | -25.0 (24.91) | -20.7 (29.71) | -15.6 (42.85)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -35.2 (38.69) | -17.2 (26.17) | -16.3 (29.29) | -7.5 (34.52)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -31.2 (34.51) | -22.9 (26.79) | -18.7 (31.17) | -6.8 (33.60)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -30.4 (33.71) | -22.4 (26.72) | -22.7 (31.60) | -2.9 (36.17)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -30.6 (29.64) | -20.6 (22.65) | -19.5 (29.54) | 0.4 (34.48)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -26.9 (28.12) | -24.7 (26.27) | -21.2 (30.95) | 3.7 (33.33)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -23.6 (26.84) | -23.8 (30.00) | -22.4 (32.85) | 4.0 (32.69)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -28.6 (33.01) | -23.0 (28.85) | -19.0 (32.29) | 8.2 (29.78)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -26.6 (34.81) | -20.2 (26.75) | -24.4 (33.78) | 6.0 (29.28)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -25.8 (32.03) | -19.7 (30.66) | -26.3 (36.36) | 8.6 (27.33)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -28.4 (32.79) | -14.7 (28.22) | -20.6 (31.61) | 6.8 (27.72)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -26.5 (32.75) | -19.0 (31.12) | -24.7 (36.95) | 8.5 (25.89)

10. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Each Visit Based on LOCF
Description: Degree of disability was self-evaluated by participant using HAQ-DI.Assessment was made based on activities capable without any aids/devices.20-question instrument assessed degree of difficulty person had in accomplishing tasks in 8 functional areas(dressing,arising,eating,walking,hygiene,reaching,gripping,and activities of daily living).Responses in each functional area were scored from 0(indicated no difficulty)to 3(indicated inability to perform task in that area).Overall score computed as: sum of domain scores and divided by number of domains answered.Total possible score range:0-3 where 0=least difficulty and 3=extreme difficulty.Data for Core Treatment Phase from Week 0-10 is reported according to participant re-randomization in 4 arms at Week 12.Data reported for Extension Phase from Baseline to Week 24,is same data for Core Treatment Phase,but excluding participants who received at least 1 dose of drug and had at least 1 postdose primary efficacy measurement after Week 24-72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
units on a scale
  Baseline | 0.90 (0.816) | 1.04 (0.770) | 0.88 (0.744) | 1.08 (0.673) | 0.85 (0.702) | 1.20 (0.789) | 0.76 (0.605) | 0.94 (0.607)
  Change at Week 2 | 0.07 (0.163) | -0.03 (0.399) | -0.08 (0.297) | 0.01 (0.258) | 0.07 (0.174) | -0.08 (0.423) | -0.04 (0.262) | 0.00 (0.270)
  Change at Week 4 | 0.03 (0.197) | -0.25 (0.460) | -0.10 (0.371) | -0.03 (0.316) | 0.02 (0.203) | -0.30 (0.485) | -0.05 (0.333) | -0.05 (0.334)
  Change at Week 8 | -0.04 (0.181) | -0.38 (0.595) | -0.10 (0.344) | -0.05 (0.404) | -0.07 (0.174) | -0.47 (0.647) | -0.09 (0.355) | -0.10 (0.428)
  Change at Week 12 | 0.12 (0.358) | -0.25 (0.357) | -0.06 (0.459) | -0.02 (0.497) | 0.10 (0.369) | -0.34 (0.340) | -0.07 (0.478) | -0.04 (0.507)
  Change at Week 16 | 0.03 (0.376) | -0.11 (0.395) | -0.11 (0.495) | -0.04 (0.421) | 0.02 (0.405) | -0.22 (0.354) | -0.13 (0.510) | -0.04 (0.457)
  Change at Week 20 | -0.04 (0.400) | -0.21 (0.341) | -0.15 (0.619) | -0.02 (0.579) | -0.07 (0.426) | -0.30 (0.341) | -0.19 (0.624) | 0.04 (0.604)
  Change at Week 24 | -0.04 (0.483) | -0.23 (0.395) | -0.23 (0.574) | 0.02 (0.464) | -0.07 (0.517) | -0.33 (0.388) | -0.28 (0.569) | 0.04 (0.510)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -0.10 (0.521) | -0.31 (0.401) | -0.25 (0.448) | 0.23 (0.770)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -0.09 (0.596) | -0.26 (0.469) | -0.13 (0.518) | 0.06 (0.461)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -0.13 (0.545) | -0.23 (0.467) | -0.18 (0.450) | 0.19 (0.409)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -0.04 (0.620) | -0.26 (0.495) | -0.16 (0.458) | 0.18 (0.457)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -0.10 (0.557) | -0.24 (0.514) | -0.18 (0.441) | 0.26 (0.488)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -0.13 (0.534) | -0.31 (0.566) | -0.18 (0.464) | 0.23 (0.432)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -0.14 (0.588) | -0.25 (0.565) | -0.21 (0.443) | 0.24 (0.370)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -0.14 (0.629) | -0.25 (0.565) | -0.19 (0.429) | 0.28 (0.362)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -0.13 (0.664) | -0.20 (0.522) | -0.12 (0.452) | 0.24 (0.370)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -0.14 (0.682) | -0.18 (0.534) | -0.16 (0.496) | 0.28 (0.471)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -0.13 (0.672) | -0.22 (0.542) | -0.17 (0.480) | 0.25 (0.391)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -0.17 (0.632) | -0.20 (0.540) | -0.15 (0.575) | 0.24 (0.473)

11. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) Values at Each Visit Based on LOCF
Description: CRP of each participants was measured as a part of blood biochemical tests. A normal CRP value is less than (<) 10 milligram per deciliter (mg/dL). A test result showing a CRP level greater than 10 mg/dL is a sign of chronic disease. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
mg/dL
  Baseline | 1.08 (1.299) | 2.50 (4.012) | 3.09 (3.186) | 1.68 (2.504) | 0.94 (1.097) | 1.83 (2.893) | 3.10 (3.316) | 0.81 (0.736)
  Change at Week 2 | 0.47 (0.795) | 0.02 (1.701) | -0.39 (1.438) | -0.13 (0.870) | 0.46 (0.855) | 0.23 (1.782) | -0.45 (1.473) | -0.11 (0.277)
  Change at Week 4 | 0.18 (0.507) | -0.63 (2.308) | -0.25 (0.938) | 0.73 (3.043) | 0.23 (0.525) | -0.01 (0.636) | -0.30 (0.957) | -0.02 (0.239)
  Change at Week 8 | -0.06 (0.579) | -0.33 (2.229) | -0.09 (1.277) | 0.43 (1.644) | 0.05 (0.389) | 0.30 (0.518) | -0.20 (1.262) | 0.07 (0.680)
  Change at Week 12 | 0.15 (0.978) | -0.44 (1.643) | 0.07 (2.524) | 0.40 (1.618) | 0.32 (0.814) | -0.18 (0.810) | 0.02 (2.618) | 0.33 (1.048)
  Change at Week 16 | 0.05 (1.090) | -0.42 (1.755) | 0.08 (1.943) | 0.63 (2.343) | 0.22 (0.965) | -0.10 (0.835) | -0.09 (1.909) | 0.28 (0.870)
  Change at Week 20 | 0.19 (1.278) | -0.41 (1.792) | 0.49 (2.713) | 0.56 (2.257) | 0.36 (1.180) | -0.10 (0.849) | 0.35 (2.771) | 0.37 (0.660)
  Change at Week 24 | 0.21 (1.144) | -0.31 (1.692) | -0.49 (2.893) | 0.47 (2.047) | 0.38 (1.004) | 0.15 (0.652) | -0.71 (2.892) | 0.65 (1.682)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | 0.42 (1.023) | 0.02 (1.301) | -0.65 (3.002) | 0.75 (1.678)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | 0.48 (1.250) | 0.09 (1.818) | -1.12 (2.881) | 0.69 (1.610)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | 0.81 (1.834) | 0.10 (1.625) | -1.16 (2.638) | 0.67 (1.516)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | 0.75 (1.825) | 0.25 (1.490) | -0.42 (1.840) | 1.01 (2.006)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | 1.08 (1.857) | 0.38 (1.459) | -0.50 (3.730) | 0.86 (1.559)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | 0.99 (1.783) | 0.21 (1.653) | -1.04 (2.757) | 0.98 (1.764)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | 0.83 (1.801) | 0.25 (1.642) | -1.16 (3.002) | 0.72 (1.430)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | 0.90 (1.859) | 0.63 (1.521) | -1.04 (3.060) | 0.67 (1.399)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | 0.80 (1.828) | 0.58 (1.405) | -1.04 (3.168) | 0.69 (1.376)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | 0.76 (1.803) | 0.47 (1.465) | -0.87 (2.213) | 0.77 (1.512)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | 1.10 (1.914) | 0.40 (1.641) | -1.10 (2.565) | 0.67 (1.462)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | 0.83 (1.791) | 0.29 (1.592) | -0.94 (3.036) | 0.97 (1.686)

12. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) Values at Each Visit Based on LOCF
Description: ESR were a type of blood test. An ESR was used to monitor the arthritis condition. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimeter per hour (mm/hr)
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
millimeter per hour (mm/hr)
  Baseline | 33.1 (19.55) | 44.4 (25.70) | 51.8 (34.26) | 35.3 (18.44) | 33.9 (19.56) | 41.2 (25.81) | 49.9 (34.91) | 32.3 (18.89)
  Change at Week 2 | 8.1 (14.36) | 0.2 (12.43) | 1.5 (11.63) | 1.5 (10.28) | 8.6 (15.37) | -1.2 (13.39) | -0.8 (8.28) | -1.9 (6.54)
  Change at Week 4 | 8.6 (14.66) | 2.1 (18.56) | -0.3 (11.56) | 1.4 (15.41) | 9.5 (15.59) | 1.5 (16.66) | -0.9 (11.77) | -4.0 (9.59)
  Change at Week 8 | 4.2 (9.53) | 5.4 (15.78) | -0.5 (17.72) | 3.9 (21.68) | 4.6 (10.21) | 3.5 (14.36) | -2.3 (17.05) | -2.6 (16.87)
  Change at Week 12 | 1.8 (10.14) | 5.1 (23.65) | -1.5 (22.06) | 6.8 (19.60) | 2.1 (10.80) | 4.7 (21.64) | -3.8 (21.06) | 4.5 (20.74)
  Change at Week 16 | 4.7 (10.64) | -3.4 (14.11) | -3.0 (23.33) | 3.0 (23.46) | 5.8 (10.90) | -3.4 (15.64) | -3.5 (24.22) | 0.8 (23.29)
  Change at Week 20 | 2.3 (12.72) | -0.4 (11.04) | 1.2 (31.07) | 6.9 (18.59) | 2.8 (13.45) | 0.6 (11.96) | -0.8 (31.33) | 2.7 (16.91)
  Change at Week 24 | 8.2 (17.51) | -2.7 (14.74) | -0.1 (33.28) | 9.3 (19.00) | 9.6 (18.32) | -2.4 (16.48) | -2.3 (33.60) | 4.5 (15.46)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | 6.5 (18.39) | -6.1 (13.12) | -5.2 (35.53) | 2.3 (21.19)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | 10.1 (19.73) | -2.5 (19.24) | -7.4 (39.76) | -0.8 (23.88)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | 10.6 (19.70) | -1.4 (20.41) | -4.1 (30.55) | -0.3 (25.25)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | 12.2 (18.88) | -3.8 (16.78) | -3.4 (19.89) | 3.0 (31.65)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | 12.2 (18.67) | 0.8 (17.87) | -4.8 (21.23) | 8.1 (26.33)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | 11.8 (18.90) | -2.5 (18.18) | -6.0 (25.17) | 5.7 (32.19)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | 16.1 (17.46) | -1.3 (18.77) | -5.6 (26.41) | 0.9 (22.43)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | 14.8 (20.93) | 1.4 (18.92) | -6.3 (28.79) | 1.2 (26.16)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | 15.2 (18.43) | 3.5 (19.91) | -5.7 (28.67) | 3.7 (25.95)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | 15.3 (17.84) | 1.0 (17.38) | -3.5 (21.04) | 3.0 (26.24)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | 16.5 (17.88) | 1.6 (20.10) | -4.6 (23.94) | 2.8 (25.88)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | 16.5 (18.00) | 3.1 (20.22) | -4.4 (26.88) | 7.1 (28.04)

13. Secondary Outcome: Change From Baseline in Disease Activity Score 28 (DAS28)-ESR Values at Each Visit Based on LOCF
Description: The DAS28 index was a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and ESR value. Total score ranged between 0-10. A DAS28-ESR score of 5.1 or above=high disease activity, a value greater than (>) 3.2 and less than or equal to (<=) 5.1=moderate disease activity and value <=3.2=low disease activity, value <2.6=disease remission. A positive change in score indicates worsening, and a negative change indicates improvement. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
score on a scale
  Baseline | 5.479 (1.2520) | 5.870 (1.3037) | 5.951 (1.1584) | 5.971 (0.9561) | 5.460 (0.9793) | 5.696 (1.3749) | 5.849 (1.1389) | 5.623 (0.5133)
  Change at Week 2 | -0.212 (0.5989) | -0.340 (0.5440) | -0.401 (0.7715) | -0.658 (0.4838) | -0.262 (0.6308) | -0.363 (0.6115) | -0.426 (0.7970) | -0.593 (0.5036)
  Change at Week 4 | -0.546 (1.1731) | -0.674 (1.0013) | -0.489 (1.0301) | -0.870 (0.7421) | -0.582 (1.2502) | -0.697 (1.0573) | -0.446 (1.0589) | -0.971 (0.7646)
  Change at Week 8 | -0.719 (0.9115) | -0.797 (1.7366) | -0.452 (1.0405) | -1.098 (0.6243) | -0.739 (0.9760) | -0.928 (1.9411) | -0.390 (1.0558) | -1.199 (0.6263)
  Change at Week 12 | -0.633 (1.1583) | -0.532 (1.4324) | -0.710 (1.2693) | -1.012 (0.8396) | -0.749 (1.1879) | -0.654 (1.5342) | -0.727 (1.3193) | -1.121 (0.8512)
  Change at Week 16 | -0.915 (1.3442) | -1.005 (0.9633) | -0.686 (1.2377) | -1.431 (0.9735) | -0.910 (1.4311) | -1.148 (1.0416) | -0.664 (1.2855) | -1.475 (0.9937)
  Change at Week 20 | -1.052 (1.2322) | -0.983 (1.0665) | -0.593 (1.4253) | -1.459 (1.1873) | -1.119 (1.3126) | -1.114 (1.1754) | -0.622 (1.4794) | -1.316 (1.0018)
  Change at Week 24 | -1.144 (1.3770) | -0.880 (1.5753) | -0.621 (1.4654) | -1.237 (1.2485) | -1.226 (1.4651) | -0.996 (1.7744) | -0.651 (1.5206) | -1.250 (1.3487)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -1.021 (1.5467) | -1.400 (1.8959) | -0.717 (1.5407) | -1.265 (1.5622)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -0.755 (1.5599) | -1.015 (1.7114) | -0.973 (2.0715) | -1.283 (1.5960)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -1.009 (1.6211) | -1.136 (1.9269) | -0.733 (1.6623) | -1.210 (1.7566)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -0.790 (1.5655) | -1.167 (1.8142) | -0.954 (1.7462) | -0.976 (1.6523)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -0.900 (1.6899) | -1.156 (2.0018) | -0.895 (1.7231) | -0.736 (1.5585)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -0.849 (1.5612) | -1.316 (2.1913) | -0.881 (1.7674) | -0.697 (1.4635)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -0.552 (1.3993) | -1.283 (2.3802) | -1.026 (1.8598) | -1.146 (1.5067)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -0.779 (1.5890) | -1.262 (2.2876) | -0.889 (1.8339) | -0.967 (1.5410)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -0.634 (1.4797) | -0.804 (1.4963) | -1.119 (2.0381) | -0.991 (1.5604)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -0.544 (1.4247) | -0.683 (1.4337) | -1.182 (2.0758) | -0.925 (1.6162)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -0.653 (1.4101) | -0.854 (1.6351) | -0.908 (2.1318) | -0.830 (1.5182)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -0.654 (1.4252) | -1.076 (1.8640) | -1.169 (2.1891) | -0.684 (1.4746)

14. Secondary Outcome: Change From Baseline in DAS28-CRP Values at Each Visit Based on LOCF
Description: The DAS28 index was a composite score of weighted components including tender joint counts of 28, swollen joint counts of 28, participant global assessment of disease activity score, and CRP value. Total score ranged between 0-10. A DAS28-CRP score of 4.1 or above=high disease activity, a value >2.7 and <=4.1=moderate disease activity and a value <=2.7=low disease activity, value <2.3=disease remission. A positive change in score indicates worsening, and a negative change indicates improvement. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
score on a scale
  Baseline | 4.842 (1.2628) | 5.194 (1.2869) | 5.305 (1.1055) | 5.318 (1.0756) | 4.780 (0.9932) | 5.033 (1.3186) | 5.218 (1.0996) | 4.909 (0.5330)
  Change at Week 2 | -0.277 (0.5794) | -0.313 (0.4086) | -0.459 (0.7658) | -0.691 (0.5431) | -0.353 (0.5823) | -0.314 (0.4634) | -0.475 (0.7948) | -0.596 (0.5478)
  Change at Week 4 | -0.672 (1.0587) | -0.653 (0.7404) | -0.550 (1.0307) | -0.808 (0.6209) | -0.719 (1.1249) | -0.607 (0.7575) | -0.510 (1.0611) | -0.881 (0.6595)
  Change at Week 8 | -0.790 (0.8574) | -0.806 (1.4652) | -0.448 (1.0170) | -1.108 (0.5967) | -0.802 (0.9214) | -0.864 (1.6578) | -0.381 (1.0262) | -1.167 (0.6389)
  Change at Week 12 | -0.567 (1.0958) | -0.559 (1.2972) | -0.704 (1.1604) | -1.095 (0.8393) | -0.657 (1.1280) | -0.680 (1.3724) | -0.710 (1.2076) | -1.196 (0.8728)
  Change at Week 16 | -1.032 (1.3230) | -0.807 (0.7085) | -0.662 (1.1490) | -1.448 (1.0766) | -1.020 (1.4086) | -0.923 (0.7435) | -0.652 (1.1953) | -1.501 (1.1190)
  Change at Week 20 | -1.086 (1.2175) | -0.913 (0.9640) | -0.569 (1.2364) | -1.501 (1.1683) | -1.152 (1.3004) | -1.054 (1.0421) | -0.595 (1.2832) | -1.329 (1.0122)
  Change at Week 24 | -1.226 (1.2308) | -0.744 (1.3057) | -0.664 (1.3388) | -1.312 (1.2535) | -1.313 (1.3047) | -0.821 (1.4747) | -0.696 (1.3878) | -1.275 (1.3575)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -1.080 (1.4327) | -1.159 (1.5168) | -0.753 (1.3526) | -1.265 (1.5105)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -0.864 (1.4813) | -0.846 (1.4961) | -1.012 (1.7898) | -1.224 (1.4763)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -1.045 (1.4527) | -1.209 (1.4589) | -0.801 (1.5149) | -1.120 (1.5781)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -0.883 (1.4812) | -1.093 (1.3147) | -0.965 (1.5133) | -0.886 (1.4063)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -0.939 (1.6417) | -1.198 (1.5077) | -0.934 (1.5769) | -0.761 (1.5076)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -0.878 (1.4321) | -1.267 (1.7114) | -0.866 (1.5055) | -0.653 (1.2861)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -0.688 (1.2532) | -1.248 (1.8622) | -1.023 (1.6672) | -1.057 (1.3742)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -0.817 (1.3728) | -1.232 (1.8140) | -0.877 (1.6018) | -0.914 (1.3941)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -0.787 (1.3827) | -0.794 (1.1386) | -1.070 (1.7630) | -0.948 (1.4326)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -0.713 (1.3495) | -0.688 (1.1425) | -1.184 (1.8181) | -0.890 (1.4800)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -0.779 (1.2602) | -0.850 (1.2527) | -0.871 (1.8144) | -0.818 (1.4112)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -0.836 (1.2718) | -1.152 (1.5226) | -1.156 (1.9211) | -0.682 (1.3581)

15. Secondary Outcome: Change From Baseline in Simple Disease Activity Index (SDAI) Values at Each Visit Based on LOCF
Description: The SDAI was calculated from tender joint counts of 28 (score range as 0-28), swollen joint counts of 28 (score range as 0-28), participant's global assessment of disease activity (score range as 0-10), physician global assessment of disease activity score (score range as 0-10), and CRP value (score range as 0-10). Total score ranged between 0-86. SDAI score of 26 or above=high disease activity, a value >11 and <=26=moderate disease activity and value <=11=low disease activity, value <=3.3=disease remission. Higher scores indicated higher disease activity. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
score on a scale
  Baseline | 29.767 (13.8824) | 34.986 (16.9418) | 33.750 (11.5847) | 34.508 (14.2748) | 28.431 (11.1731) | 33.745 (17.7674) | 33.069 (11.7626) | 29.060 (6.6750)
  Change at Week 2 | -5.620 (7.5960) | -5.607 (7.1229) | -6.100 (9.3523) | -9.075 (8.0323) | -6.054 (8.1006) | -5.873 (8.0467) | -6.362 (9.6807) | -6.640 (6.2285)
  Change at Week 4 | -7.767 (9.6279) | -10.221 (11.8874) | -6.836 (12.3932) | -9.667 (5.8116) | -8.062 (10.2120) | -9.382 (11.9577) | -6.392 (12.7832) | -9.790 (6.4160)
  Change at Week 8 | -10.260 (8.9168) | -11.136 (18.0780) | -5.586 (13.8352) | -13.008 (5.7949) | -10.023 (9.5951) | -11.545 (20.3240) | -4.985 (14.2086) | -12.930 (6.3990)
  Change at Week 12 | -6.793 (10.2078) | -8.421 (17.5072) | -7.643 (14.2285) | -12.792 (8.4873) | -9.023 (12.2819) | -9.827 (18.8785) | -7.815 (14.7942) | -13.080 (9.0454)
  Change at Week 16 | -11.760 (13.4649) | -12.700 (11.1552) | -8.521 (14.8650) | -14.917 (10.6017) | -11.762 (14.5004) | -13.809 (12.3841) | -8.446 (15.4692) | -14.290 (10.4209)
  Change at Week 20 | -12.167 (14.0241) | -13.536 (13.7755) | -6.907 (15.9803) | -17.033 (11.3561) | -12.708 (15.0684) | -14.964 (15.3173) | -7.285 (16.5677) | -14.760 (8.8873)
  Change at Week 24 | -14.107 (13.4448) | -12.086 (16.8719) | -7.171 (16.5184) | -13.517 (12.9978) | -14.946 (14.3229) | -13.109 (19.0562) | -7.569 (17.1230) | -11.670 (12.9570)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -13.708 (15.3680) | -13.945 (20.3219) | -7.954 (17.7855) | -11.230 (13.3073)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -12.169 (15.7365) | -11.855 (18.5106) | -8.708 (19.9022) | -10.890 (14.0719)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -12.569 (15.7788) | -14.655 (19.3982) | -8.600 (19.1369) | -9.300 (17.4237)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -11.438 (15.7793) | -13.945 (18.4699) | -10.215 (17.5279) | -7.950 (17.2220)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -11.277 (17.4198) | -14.509 (19.4841) | -9.285 (19.7611) | -6.820 (16.7918)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -11.685 (15.4954) | -15.073 (20.5706) | -9.731 (19.3009) | -5.180 (14.7420)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -8.469 (13.4793) | -14.682 (22.2529) | -10.369 (20.2755) | -8.480 (15.8229)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -9.577 (14.5219) | -14.700 (21.6976) | -9.177 (19.7402) | -7.060 (15.2876)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -9.269 (14.6406) | -11.373 (16.1736) | -10.915 (20.8181) | -7.780 (16.2905)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -8.677 (14.0686) | -9.055 (15.1680) | -10.831 (20.7975) | -6.600 (16.3039)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -9.077 (13.8200) | -10.527 (18.0938) | -9.054 (20.5279) | -6.240 (15.4074)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -9.122 (13.6836) | -12.956 (19.9469) | -10.985 (21.6004) | -5.359 (15.1614)

16. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Values at Each Visit Based on LOCF
Description: The CDAI was calculated from tender joint counts of 28 (score range as 0-28), swollen joint counts of 28 (score range as 0-28), participant's global assessment of disease activity (score range as 0-10) and physician global assessment of disease activity (score range as 0-10). Total score ranged between 0-76. CDAI score of 22 or above=high disease activity, a value >10 and <=22=moderate disease activity, a value <=10=low disease activity, and a value <=2.8=disease remission. Higher scores indicated higher disease activity. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Baseline to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
score on a scale
  Baseline | 28.687 (13.2790) | 32.486 (15.4890) | 30.657 (9.4928) | 32.833 (12.8294) | 27.492 (11.0621) | 31.918 (17.1251) | 29.969 (9.5103) | 28.250 (6.6991)
  Change at Week 2 | -6.087 (7.2870) | -5.629 (6.6070) | -5.714 (9.0823) | -8.942 (8.1025) | -6.515 (7.7685) | -6.100 (7.3778) | -5.908 (9.4231) | -6.530 (6.2243)
  Change at Week 4 | -7.947 (9.5817) | -9.593 (11.0959) | -6.586 (12.2036) | -10.400 (6.4684) | -8.292 (10.1373) | -9.373 (11.9883) | -6.092 (12.5557) | -9.770 (6.4534)
  Change at Week 8 | -10.200 (9.0094) | -10.807 (18.0182) | -5.493 (13.6155) | -13.433 (5.8262) | -10.077 (9.6871) | -11.845 (20.2785) | -4.785 (13.9004) | -13.000 (6.1248)
  Change at Week 12 | -8.653 (11.3262) | -7.986 (17.5102) | -7.714 (12.9650) | -13.192 (8.6300) | -9.438 (11.8829) | -9.645 (19.0353) | -7.831 (13.4867) | -13.410 (8.7252)
  Change at Week 16 | -11.807 (12.8912) | -12.279 (11.3618) | -8.600 (13.6702) | -15.550 (11.7076) | -11.985 (13.8258) | -13.709 (12.4778) | -8.354 (14.1961) | -14.570 (10.3295)
  Change at Week 20 | -12.360 (13.3098) | -13.129 (14.0345) | -7.400 (14.5217) | -17.592 (12.6565) | -13.069 (14.2281) | -14.864 (15.4843) | -7.638 (15.0861) | -15.130 (8.6208)
  Change at Week 24 | -14.320 (12.8371) | -11.779 (16.9787) | -6.679 (14.8931) | -13.983 (12.3963) | -15.331 (13.5575) | -13.255 (19.0433) | -6.862 (15.4849) | -12.320 (11.8315)
  Change at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 28 |  |  |  |  | -14.123 (14.6710) | -13.964 (20.1448) | -7.300 (15.9008) | -11.980 (12.1211)
  Change at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 32 |  |  |  |  | -12.646 (14.8310) | -11.945 (18.0326) | -7.585 (17.9281) | -11.580 (12.9276)
  Change at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 36 |  |  |  |  | -13.377 (14.4734) | -14.755 (19.2637) | -7.438 (17.2899) | -9.970 (16.6191)
  Change at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 40 |  |  |  |  | -12.192 (14.5243) | -14.200 (18.3184) | -9.792 (17.3534) | -8.960 (16.2228)
  Change at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 44 |  |  |  |  | -12.354 (16.1397) | -14.891 (19.2430) | -8.785 (18.0594) | -7.680 (16.0389)
  Change at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 48 |  |  |  |  | -12.677 (14.3445) | -15.282 (20.3093) | -8.692 (17.4611) | -6.160 (14.0400)
  Change at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 52 |  |  |  |  | -9.300 (12.3597) | -14.936 (21.9162) | -9.208 (18.0779) | -9.200 (15.1983)
  Change at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 56 |  |  |  |  | -10.823 (13.4309) | -15.327 (21.3345) | -8.138 (17.6150) | -7.730 (14.7041)
  Change at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 60 |  |  |  |  | -10.415 (13.4300) | -11.955 (15.8809) | -9.877 (18.6515) | -8.470 (15.7053)
  Change at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 64 |  |  |  |  | -9.785 (12.9341) | -9.527 (14.8393) | -9.962 (19.4745) | -7.370 (15.5947)
  Change at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 68 |  |  |  |  | -10.523 (12.9377) | -10.927 (17.8324) | -7.954 (18.5732) | -6.910 (14.6880)
  Change at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Change at Week 72 |  |  |  |  | -10.300 (12.7026) | -13.245 (19.5791) | -10.046 (19.5472) | -6.330 (14.3787)

17. Secondary Outcome: Number of Participants With a European League Against Rheumatism (EULAR) Good, Moderate or No Response Using DAS28-ESR at Each Visit Based on NRI
Description: The Disease Activity Score Based on 28-joints Count-ESR based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 <=3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to <=5.1 or change from baseline >0.6 to <=1.2 with DAS28 <=5.1; non-responders: change from baseline <=0.6 or change from baseline >0.6 and <=1.2 with DAS28 >5.1. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
Participants
  EULAR Response at Week 2: Good Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EULAR Response at Week 2: Moderate Response | 2 | 4 | 4 | 4 | 2 | 4 | 4 | 4
  EULAR Response at Week 2: No Response | 13 | 10 | 10 | 8 | 11 | 7 | 9 | 6
  EULAR Response at Week 4: Good Response | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 0
  EULAR Response at Week 4: Moderate Response | 3 | 4 | 4 | 5 | 2 | 3 | 4 | 5
  EULAR Response at Week 4: No Response | 10 | 10 | 9 | 7 | 9 | 8 | 8 | 5
  EULAR Response at Week 8: Good Response | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  EULAR Response at Week 8: Moderate Response | 4 | 5 | 5 | 7 | 3 | 4 | 4 | 7
  EULAR Response at Week 8: No Response | 10 | 8 | 9 | 5 | 9 | 6 | 9 | 3
  EULAR Response at Week 12: Good Response | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 0
  EULAR Response at Week 12: Moderate Response | 5 | 4 | 5 | 7 | 5 | 3 | 5 | 7
  EULAR Response at Week 12: No Response | 9 | 10 | 7 | 5 | 7 | 8 | 6 | 3
  EULAR Response at Week 16: Good Response | 3 | 0 | 1 | 2 | 2 | 0 | 1 | 2
  EULAR Response at Week 16: Moderate Response | 5 | 6 | 5 | 5 | 5 | 5 | 5 | 4
  EULAR Response at Week 16: No Response | 7 | 8 | 8 | 5 | 6 | 6 | 7 | 4
  EULAR Response at Week 20: Good Response | 3 | 1 | 2 | 2 | 3 | 1 | 2 | 2
  EULAR Response at Week 20: Moderate Response | 8 | 6 | 4 | 5 | 7 | 5 | 4 | 4
  EULAR Response at Week 20: No Response | 4 | 7 | 8 | 5 | 3 | 5 | 7 | 4
  EULAR Response at Week 24: Good Response | 2 | 2 | 1 | 2 | 2 | 2 | 1 | 2
  EULAR Response at Week 24: Moderate Response | 8 | 2 | 5 | 6 | 8 | 2 | 5 | 5
  EULAR Response at Week 24: No Response | 5 | 10 | 8 | 4 | 3 | 7 | 7 | 3
  EULAR Response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 28: Good Response |  |  |  |  | 1 | 4 | 2 | 3
  EULAR Response at Week 28: Moderate Response |  |  |  |  | 8 | 3 | 4 | 3
  EULAR Response at Week 28: No Response |  |  |  |  | 4 | 4 | 7 | 4
  EULAR Response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 32: Good Response |  |  |  |  | 1 | 2 | 3 | 3
  EULAR Response at Week 32: Moderate Response |  |  |  |  | 5 | 3 | 1 | 4
  EULAR Response at Week 32: No Response |  |  |  |  | 7 | 6 | 9 | 3
  EULAR Response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 36: Good Response |  |  |  |  | 2 | 3 | 1 | 3
  EULAR Response at Week 36: Moderate Response |  |  |  |  | 8 | 2 | 5 | 4
  EULAR Response at Week 36: No Response |  |  |  |  | 3 | 6 | 7 | 3
  EULAR Response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 40: Good Response |  |  |  |  | 3 | 5 | 2 | 1
  EULAR Response at Week 40: Moderate Response |  |  |  |  | 5 | 0 | 5 | 4
  EULAR Response at Week 40: No Response |  |  |  |  | 5 | 6 | 6 | 5
  EULAR Response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 44: Good Response |  |  |  |  | 2 | 4 | 1 | 1
  EULAR Response at Week 44: Moderate Response |  |  |  |  | 6 | 1 | 5 | 5
  EULAR Response at Week 44: No Response |  |  |  |  | 5 | 6 | 7 | 4
  EULAR Response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 48: Good Response |  |  |  |  | 1 | 4 | 3 | 1
  EULAR Response at Week 48: Moderate Response |  |  |  |  | 8 | 2 | 2 | 4
  EULAR Response at Week 48: No Response |  |  |  |  | 4 | 5 | 8 | 5
  EULAR Response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 52: Good Response |  |  |  |  | 1 | 4 | 3 | 1
  EULAR Response at Week 52: Moderate Response |  |  |  |  | 6 | 2 | 3 | 6
  EULAR Response at Week 52: No Response |  |  |  |  | 6 | 5 | 7 | 3
  EULAR Response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 56: Good Response |  |  |  |  | 2 | 3 | 3 | 1
  EULAR Response at Week 56: Moderate Response |  |  |  |  | 6 | 3 | 2 | 3
  EULAR Response at Week 56: No Response |  |  |  |  | 5 | 5 | 8 | 6
  EULAR Response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 60: Good Response |  |  |  |  | 1 | 3 | 3 | 2
  EULAR Response at Week 60: Moderate Response |  |  |  |  | 7 | 2 | 3 | 3
  EULAR Response at Week 60: No Response |  |  |  |  | 5 | 6 | 7 | 5
  EULAR Response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 64: Good Response |  |  |  |  | 1 | 3 | 2 | 2
  EULAR Response at Week 64: Moderate Response |  |  |  |  | 6 | 2 | 4 | 1
  EULAR Response at Week 64: No Response |  |  |  |  | 6 | 6 | 7 | 7
  EULAR Response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 68: Good Response |  |  |  |  | 0 | 2 | 1 | 1
  EULAR Response at Week 68: Moderate Response |  |  |  |  | 7 | 4 | 4 | 2
  EULAR Response at Week 68: No Response |  |  |  |  | 6 | 5 | 8 | 7
  EULAR Response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR Response at Week 72: Good Response |  |  |  |  | 1 | 2 | 3 | 1
  EULAR Response at Week 72: Moderate Response |  |  |  |  | 5 | 4 | 2 | 2
  EULAR Response at Week 72: No Response |  |  |  |  | 7 | 5 | 8 | 7

18. Secondary Outcome: Number of Participants With a EULAR Good, Moderate or No Response Using DAS28-CRP at Each Visit Based on NRI
Description: The Disease Activity Score Based on 28-joints Count-CRP based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 <=3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to <=5.1 or change from baseline >0.6 to <=1.2 with DAS28 <=5.1; non-responders: change from baseline <=0.6 or change from baseline >0.6 and <=1.2 with DAS28 >5.1. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
Participants
  EULAR response at Week 2: Good response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EULAR response at Week 2: Moderate response | 1 | 1 | 3 | 4 | 1 | 1 | 3 | 3
  EULAR response at Week 2: No response | 14 | 13 | 11 | 8 | 12 | 10 | 10 | 7
  EULAR response at Week 4: Good response | 2 | 0 | 1 | 1 | 2 | 0 | 1 | 1
  EULAR response at Week 4: Moderate response | 3 | 4 | 3 | 4 | 2 | 3 | 3 | 4
  EULAR response at Week 4: No response | 10 | 10 | 10 | 7 | 9 | 8 | 9 | 5
  EULAR response at Week 8: Good response | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1
  EULAR response at Week 8: Moderate response | 6 | 4 | 5 | 6 | 5 | 3 | 4 | 6
  EULAR response at Week 8: No response | 9 | 9 | 9 | 5 | 8 | 7 | 9 | 3
  EULAR response at Week 12: Good response | 1 | 0 | 2 | 3 | 1 | 0 | 2 | 3
  EULAR response at Week 12: Moderate response | 4 | 4 | 3 | 3 | 4 | 3 | 3 | 3
  EULAR response at Week 12: No response | 10 | 10 | 9 | 6 | 8 | 8 | 8 | 4
  EULAR response at Week 16: Good response | 3 | 1 | 2 | 4 | 2 | 1 | 2 | 4
  EULAR response at Week 16: Moderate response | 6 | 4 | 4 | 3 | 6 | 3 | 4 | 2
  EULAR response at Week 16: No response | 6 | 9 | 8 | 5 | 5 | 7 | 7 | 4
  EULAR response at Week 20: Good response | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 3
  EULAR response at Week 20: Moderate response | 9 | 5 | 3 | 4 | 8 | 4 | 3 | 3
  EULAR response at Week 20: No response | 4 | 7 | 9 | 5 | 3 | 5 | 8 | 4
  EULAR response at Week 24: Good response | 3 | 1 | 1 | 4 | 3 | 1 | 1 | 4
  EULAR response at Week 24: Moderate response | 8 | 3 | 4 | 4 | 8 | 3 | 4 | 3
  EULAR response at Week 24: No response | 4 | 10 | 9 | 4 | 2 | 7 | 8 | 3
  EULAR response at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 28: Good response |  |  |  |  | 1 | 3 | 2 | 4
  EULAR response at Week 28: Moderate response |  |  |  |  | 9 | 3 | 4 | 2
  EULAR response at Week 28: No response |  |  |  |  | 3 | 5 | 7 | 4
  EULAR response at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 32: Good response |  |  |  |  | 1 | 3 | 3 | 3
  EULAR response at Week 32: Moderate response |  |  |  |  | 7 | 2 | 2 | 4
  EULAR response at Week 32: No response |  |  |  |  | 5 | 6 | 8 | 3
  EULAR response at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 36: Good response |  |  |  |  | 3 | 4 | 1 | 3
  EULAR response at Week 36: Moderate response |  |  |  |  | 7 | 2 | 4 | 4
  EULAR response at Week 36: No response |  |  |  |  | 3 | 5 | 8 | 3
  EULAR response at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 40: Good response |  |  |  |  | 2 | 1 | 2 | 2
  EULAR response at Week 40: Moderate response |  |  |  |  | 5 | 4 | 3 | 4
  EULAR response at Week 40: No response |  |  |  |  | 6 | 6 | 8 | 4
  EULAR response at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 44: Good response |  |  |  |  | 3 | 4 | 2 | 2
  EULAR response at Week 44: Moderate response |  |  |  |  | 5 | 1 | 4 | 3
  EULAR response at Week 44: No response |  |  |  |  | 5 | 6 | 7 | 5
  EULAR response at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 48: Good response |  |  |  |  | 1 | 3 | 2 | 1
  EULAR response at Week 48: Moderate response |  |  |  |  | 6 | 3 | 3 | 4
  EULAR response at Week 48: No response |  |  |  |  | 6 | 5 | 8 | 5
  EULAR response at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 52: Good response |  |  |  |  | 1 | 3 | 2 | 1
  EULAR response at Week 52: Moderate response |  |  |  |  | 6 | 3 | 4 | 6
  EULAR response at Week 52: No response |  |  |  |  | 6 | 5 | 7 | 3
  EULAR response at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 56: Good response |  |  |  |  | 2 | 3 | 2 | 1
  EULAR response at Week 56: Moderate response |  |  |  |  | 6 | 3 | 2 | 3
  EULAR response at Week 56: No response |  |  |  |  | 5 | 5 | 9 | 6
  EULAR response at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 60: Good response |  |  |  |  | 2 | 2 | 2 | 2
  EULAR response at Week 60: Moderate response |  |  |  |  | 5 | 3 | 3 | 3
  EULAR response at Week 60: No response |  |  |  |  | 6 | 6 | 8 | 5
  EULAR response at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 64: Good response |  |  |  |  | 2 | 2 | 3 | 2
  EULAR response at Week 64: Moderate response |  |  |  |  | 4 | 2 | 4 | 2
  EULAR response at Week 64: No response |  |  |  |  | 7 | 7 | 6 | 6
  EULAR response at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 68: Good response |  |  |  |  | 1 | 2 | 2 | 2
  EULAR response at Week 68: Moderate response |  |  |  |  | 6 | 4 | 3 | 1
  EULAR response at Week 68: No response |  |  |  |  | 6 | 5 | 8 | 7
  EULAR response at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  EULAR response at Week 72: Good response |  |  |  |  | 2 | 3 | 3 | 1
  EULAR response at Week 72: Moderate response |  |  |  |  | 3 | 3 | 3 | 2
  EULAR response at Week 72: No response |  |  |  |  | 8 | 5 | 7 | 7

19. Secondary Outcome: Percentage of Participants Who Achieved SDAI Remission at Each Visit Based on NRI
Description: The SDAI was calculated from tender joint counts of 28 (score range as 0-28), swollen joint counts of 28 (score range as 0-28), participant's global assessment of disease activity (score range as 0-10), physician global assessment of disease activity score (score range as 0-10), and CRP value (score range as 0-10). Total score ranged between 0-86. SDAI score of 86 or above=high disease activity, a value >11 and <=26=moderate disease activity, a value >=3.4 and <=11=low disease activity. Higher scores indicated higher disease activity. SDAI Remission was defined as SDAI score <=3.3. Data for Core Treatment Phase from Week 0-10 is reported according to participant's re-randomization in four arms at Week 12. Data reported for Extension Phase from Week 2 to Week 24, is same data for Core Treatment Phase, but excluding participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
percentage of participants
  Remission at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 4 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Remission at Week 8 | 6.7 [0.00 to 19.29] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 12 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Remission at Week 16 | 6.7 [0.00 to 19.29] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 8.3 [0.00 to 23.97] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 20 | 6.7 [0.00 to 19.29] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 8.3 [0.00 to 23.97] | 7.7 [0.00 to 22.18] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 24 | 6.7 [0.00 to 19.29] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 8.3 [0.00 to 23.97] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 28 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Remission at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 32 |  |  |  |  | 7.7 [0.00 to 22.18] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 36 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 40 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 44 |  |  |  |  | 7.7 [0.00 to 22.18] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 48 |  |  |  |  | 7.7 [0.00 to 22.18] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 52 |  |  |  |  | 0.0 [0.00 to 0.00] | 27.3 [0.95 to 53.59] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 56 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 60 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 64 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 68 |  |  |  |  | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 72 |  |  |  |  | 0.0 [0.00 to 0.00] | 27.3 [0.95 to 53.59] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]

20. Secondary Outcome: Percentage of Participants Who Achieved CDAI Remission at Each Visit Based on NRI
Description: The CDAI was calculated from tender joint counts of 28 (score range as 0-28), swollen joint counts of 28 (score range as 0-28), participant's global assessment of disease activity (score range as 0-10), and physician global assessment of disease activity score (score range as 0-10). Total score ranged between 0-76. CDAI score of 76 or above=high disease activity, a value >10 and <=22=moderate disease activity, a value >2.9 and <=10=low disease activity. Higher scores indicated higher disease activity. CDAI Remission was defined as CDAI score <=2.8. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
percentage of participants
  Remission at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 4 | 6.7 [0.00 to 19.29] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 8 | 6.7 [0.00 to 19.29] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 12 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Remission at Week 16 | 6.7 [0.00 to 19.29] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 20 | 6.7 [0.00 to 19.29] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 8.3 [0.00 to 23.97] | 7.7 [0.00 to 22.18] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 24 | 6.7 [0.00 to 19.29] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 8.3 [0.00 to 23.97] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 28 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 20.0 [0.00 to 44.79]
  Remission at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 32 |  |  |  |  | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 36 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 40 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 44 |  |  |  |  | 7.7 [0.00 to 22.18] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 48 |  |  |  |  | 7.7 [0.00 to 22.18] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 52 |  |  |  |  | 0.0 [0.00 to 0.00] | 27.3 [0.95 to 53.59] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 56 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 60 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 64 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 68 |  |  |  |  | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 72 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]

21. Secondary Outcome: Percentage of Participants Who Achieved Boolean Remission at Each Visit Based on NRI
Description: Boolean remission criteria was defined as: tender joint count 68 <=1; swollen joint count 66 <=1; CRP <=1 mg/dL; and disease activity assessments VAS (mm) by participants <=10. Data for the Core Treatment Phase from Week 0-10 is reported according to the participant's re-randomization in four arms at Week 12. Data reported for the Extension Phase from Week 2 to Week 24, is the same data for the Core Treatment Phase, but excluding the participants who received at least 1 dose of study drug after Week 24 and had at least 1 postdose primary efficacy measurement after Week 24 to Week 72.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
Number analyzed (Participants) | 15 | 14 | 14 | 12 | 13 | 11 | 13 | 10
percentage of participants
  Remission at Week 2 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 4 | 6.7 [0.00 to 19.29] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 8 | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 12 | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Remission at Week 16 | 6.7 [0.00 to 19.29] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00]
  Remission at Week 20 | 13.3 [0.00 to 30.54] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 8.3 [0.00 to 23.97] | 15.4 [0.00 to 35.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 24 | 6.7 [0.00 to 19.29] | 0.0 [0.00 to 0.00] | 7.1 [0.00 to 20.63] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Remission at Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 28 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 32 |  |  |  |  | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 7.7 [0.00 to 22.18] | 0.0 [0.00 to 0.00]
  Remission at Week 36: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 36 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 40 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 44 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 48: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 48 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 52: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 52 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 7.7 [0.00 to 22.18] | 10.0 [0.00 to 28.59]
  Remission at Week 56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 56 |  |  |  |  | 0.0 [0.00 to 0.00] | 18.2 [0.00 to 40.97] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 60: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 60 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 64: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 64 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]
  Remission at Week 68: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 68 |  |  |  |  | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 0.0 [0.00 to 0.00] | 10.0 [0.00 to 28.59]
  Remission at Week 72: number analyzed (Participants) | 0 | 0 | 0 | 0 | 13 | 11 | 13 | 10
  Remission at Week 72 |  |  |  |  | 0.0 [0.00 to 0.00] | 9.1 [0.00 to 26.08] | 15.4 [0.00 to 35.00] | 10.0 [0.00 to 28.59]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 104 Weeks (Treatment Phase: From the first dose of study drug till Week 24; Extension Phase: Post Week 24 till Week 104)
Description: SAS included participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Arm/Group | Core Treatment Phase: Placebo | Core Treatment Phase: E6011 400 mg | Core Treatment Phase: Placebo Then E6011 200 mg | Core Treatment Phase: Placebo Then E6011 400 mg | Core Treatment Phase: E6011 400 mg Then E6011 200 mg | Core Treatment Phase: E6011 400 mg Then E6011 400 mg | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31 | 0/15 | 0/14 | 0/14 | 0/12 | 1/13 | 0/11 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/31 | 0/15 | 1/14 | 0/14 | 0/12 | 2/13 | 2/11 | 2/13 | 0/10
Other Adverse Events (participants affected / at risk) | 19/33 | 14/31 | 12/15 | 13/14 | 13/14 | 9/12 | 13/13 | 11/11 | 13/13 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Phase: Placebo (N=33) | Core Treatment Phase: E6011 400 mg (N=31) | Core Treatment Phase: Placebo Then E6011 200 mg (N=15) | Core Treatment Phase: Placebo Then E6011 400 mg (N=14) | Core Treatment Phase: E6011 400 mg Then E6011 200 mg (N=14) | Core Treatment Phase: E6011 400 mg Then E6011 400 mg (N=12) | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg (N=13) | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg (N=11) | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg (N=13) | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg (N=10)
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Treatment Phase: Placebo (N=33) | Core Treatment Phase: E6011 400 mg (N=31) | Core Treatment Phase: Placebo Then E6011 200 mg (N=15) | Core Treatment Phase: Placebo Then E6011 400 mg (N=14) | Core Treatment Phase: E6011 400 mg Then E6011 200 mg (N=14) | Core Treatment Phase: E6011 400 mg Then E6011 400 mg (N=12) | Extension Phase: Placebo Then E6011 200 mg Then E6011 200 mg (N=13) | Extension Phase: Placebo Then E6011 400 mg Then E6011 200 mg (N=11) | Extension Phase: E6011 400 mg Then E6011 200 mg Then E6011 200 mg (N=13) | Extension Phase: E6011 400 mg Then E6011 400 mg Then E6011 200 mg (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eustachian tube patulous (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 0
Injection site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Injection site warmth (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 3
Breast abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cell marker increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 2 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 9 | 4 | 2 | 4 | 4 | 4 | 7 | 4 | 8 | 5
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Chloasma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Poor peripheral circulation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2019-03-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT02960490/Prot_000.pdf
  • Statistical Analysis Plan: Core and Entire Treatment Phase (2018-06-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT02960490/SAP_001.pdf
  • Statistical Analysis Plan: Extension Phase (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/90/NCT02960490/SAP_002.pdf